CLINICAL TRIAL: NCT01293526
Title: Acute Optimization of Cardiac Resynchronization Therapy (CRT) Using Echocardiography and SonR
Brief Title: Acute Optimization of Cardiac Resynchronization Therapy (CRT)Using Echocardiography and SonR
Acronym: SonR Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution, no replacement
Sponsor: Piedmont Healthcare (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SonR Access
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
Keywords: Heart failure; echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental 1 (Experimental): Patients who respond will have their leads placed based on study measurements.
  Interventions: Device: Experimental
- Control (Experimental): Leads will be placed using standard procedures.
  Interventions: Device: Control
- Experimental 2 (Experimental): Patients who respond will have their leads placed based on standard lead placement.
  Interventions: Device: Experimental 2

INTERVENTIONS:
Device: Control — Patients who respond will have leads will be placed using standard procedures.
  Arms: Control
Device: Experimental — Patients who respond will have their leads placed based on study measurements.
  Arms: Experimental 1
Device: Experimental 2 — Patients who respond will have their leads placed based on standard lead placement.
  Arms: Experimental 2

SUMMARY:
The purpose of this study is to correlate the three lead placement (wires that go to the heart) possibilities and the responses from the patient's heart. This will be done with the help of an echocardiography and SonR signals, which is an external device that is capable of detecting sounds created by the heart.

DETAILED DESCRIPTION:
A cardiac resynchronization therapy defibrillator (CRT-D) is a device designed to automatically recognize and stop rapid, harmful heart beats and allow the heart to return to a safe, regular heart rhythm. The CRT-D device may help the heart pump more efficiently by improving the timing of different parts of the heart beat. A CRT-D device has three leads (wires that go to the heart). One lead is placed in one of the top chambers of the heart (right atrium), another lead is placed in the lower right chamber (right ventricle) and the third lead is placed along the side of the left ventricle. The top chambers are stimulated first, either by the natural heartbeat or by the CRT-D device if the heartbeat is too slow. Shortly after that, the bottom chambers are stimulated. By pacing the heart in this way, the doctor hopes to improve the timing of different components of the heart beat in order to improve the efficiency of the heart and to improve the patient's heart failure symptoms. The purpose of this study is to correlate the three lead placement possibilities and the responses from the patient's heart. This will be done with the help of an echocardiography and SonR signals, which is an external device that is capable of detecting sounds created by the heart.

Based on the CRT implant, special measurements will be made to optimize the placements of the device leads. Based on the success of those measurements and a patient's own response, the patient will be placed into one of three groups.

Group 1: Patients with no response

Patients with a successful response will be randomized to:

Group 2: Lead placement based on study measurements

OR

Group 3: Standard lead placement

ELIGIBILITY:
Inclusion Criteria:

* Must have been indicated for implantation or upgrade to a CRT-D system in the last 3 months
* Indicated for CRT according to current guidelines
* QRS Duration between 120 ms and 150 ms
* Able and willing to provide consent and Authorization of Use of PHI

Exclusion Criteria:

* Myocardial infarction or acute coronary syndrome deemed inappropriate for trial per the investigator within 90 days of implant
* Planned, or recent heart surgery or revascularization within the last three months
* Already enrolled in other study that precludes enrollment in this study per Principal Investigator
* Known Pregnancy at the time of enrollment
* Age less than 18 at the time of enrollment
* Unable to comply with follow-up requirements
* Chronic Atrial Fibrillation
* Recent history of medical non-compliance as determined by the investigator
* Unable or unwilling to provide consent and Authorization of Use of PHI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percent of responding patients | 6 months
  Percent of patients who have a positive response to implantation of the CRT at 6 months post-implant.

SECONDARY OUTCOMES:
Comparison of echocardiography and SonR signals | 6 months
  Correlation of the results of optimization performed by echocardiography with the optimal setting as defined by the SonR signal.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Dan, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States